CLINICAL TRIAL: NCT00272311
Title: A Randomized, Double-Blind Trial to Test Higher- Versus Lower-Doses of Aspirin on Inflammatory Markers and Platelet Biomarkers and Nitric Oxide Formation in High Risk Primary Prevention (Patients With Metabolic Syndrome)
Brief Title: Aspirin Dose and Atherosclerosis in Patients With Metabolic Syndrome
Acronym: PAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Florida Atlantic University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H08-35
Record Dates: First submitted 2006-01-03; First posted 2006-01-05 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Cardiovascular Diseases; Metabolic Syndrome X; Atherosclerosis
Keywords: Primary prevention; Cardiovascular diseases; Aspirin; Metabolic Syndrome X; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome; Atherosclerosis | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Active Comparator): 81 mg Aspirin
  Interventions: Drug: Aspirin
- 2 (Active Comparator): 162 mg Aspirin
  Interventions: Drug: Aspirin
- 3 (Active Comparator): 325 mg Aspirin
  Interventions: Drug: Aspirin
- 4 (Active Comparator): 650 mg Aspirin
  Interventions: Drug: Aspirin
- 5 (Active Comparator): 1300 mg Aspirin
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Dosage

SUMMARY:
The purpose of the study is to test higher versus lower doses of aspirin on markers of atherosclerosis in patients at risk of a first heart attack.

DETAILED DESCRIPTION:
Aspirin reduces risks of heart attacks, strokes, and deaths from cardiovascular causes in patients who have survived a prior event as well as during an acute heart attack. Aspirin also prevents a first heart attack.

Low dose aspirin is sufficient to achieve complete inhibition of platelet aggregability, or stickiness, and this is the mechanism whereby aspirin prevents formation of blood clots.

Our research is designed to explore whether higher doses of aspirin provide additional benefits on markers of atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 40 to 80 years, inclusive.

  2. No previous heart attack or a stroke, or other forms of these diseases.

  3. Have at least three of the five characteristics listed below, indicating presence of metabolic syndrome, as defined by NCEP-III:
  1. waist measuring more than 40 inches (for men) or more than 35 inches (for women),
  2. high density lipoprotein (HDL) cholesterol levels lower than 40 milligrams per deciliter (mg/dl) in men or 50 mg/dl in women,
  3. triglyceride (TG) levels above 150 mg/dl,
  4. blood pressure greater than 130 millimeters of mercury (mmHg) systolic or 85 mmHg diastolic,
  5. fasting blood sugar greater than 110 mg/dl

Exclusion Criteria:

1. Patients taking greater than 81mg aspirin daily.
2. Patients taking anti-platelet drugs such as clopidogrel or non-steroidal anti-inflammatory drugs (NSAIDs) or anticoagulant drugs such as warfarin, during the last two weeks.
3. Patients taking any of the following medications for less than 3 months, or who plan to take them for the first time during the next 3 months: ACE-inhibitors, angiotensin receptor blockers, calcium channel blockers, or statins.
4. Patients who are currently cigarette smokers.
5. Women patients who are pregnant, planning to become pregnant, nursing a child, or taking hormone replacement therapy.
6. Patients with any coagulation, bleeding or blood disorders.
7. Patients who are sensitive or allergic to aspirin.
8. Patients with documented history of any gastrointestinal disorders, including bleeding ulcers.
9. Patients with any evidence of cancer or history of significant cardiovascular disease (including heart attack, stroke or drop attacks termed transient ischemic attacks (TIAs), or blockages of the arteries in the legs termed peripheral arterial disease (PAD)), kidney, liver, lung, blood, or brain disorders.
10. Patients with asthma, rhinitis, or nasal polyps.
11. Patients with any abnormal laboratory value or physical finding that, in the view of the responsible clinician, may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety.
12. Patients with Class IV heart failure.
13. Patients with severe aortic insufficiency, or aortic regurgitation.
14. Patients with hearing loss or tinnitus.
15. Patients with tremors which cause them not to be able to remain motionless for approximately 30 seconds.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Hennekens, MD, DrPH, Principal Investigator — Florida Atlantic University; Wendy R Schneider, MSN, CCRC, Study Director — Florida Atlantic University
Locations (1):
- HeartDrug Research, LLC, Towson, Maryland, United States

REFERENCES:
- [Background] Williams A, Hennekens CH. The role of aspirin in cardiovascular diseases--forgotten benefits? Expert Opin Pharmacother. 2004 Jan;5(1):109-15. doi: 10.1517/14656566.5.1.109. PMID 14680440
- [Background] Hennekens CH, Buring JE, Sandercock P, Collins R, Peto R. Aspirin and other antiplatelet agents in the secondary and primary prevention of cardiovascular disease. Circulation. 1989 Oct;80(4):749-56. doi: 10.1161/01.cir.80.4.749. No abstract available. PMID 2676237
- [Background] Eidelman RS, Hebert PR, Weisman SM, Hennekens CH. An update on aspirin in the primary prevention of cardiovascular disease. Arch Intern Med. 2003 Sep 22;163(17):2006-10. doi: 10.1001/archinte.163.17.2006. PMID 14504112
- [Background] Roth GJ, Stanford N, Majerus PW. Acetylation of prostaglandin synthase by aspirin. Proc Natl Acad Sci U S A. 1975 Aug;72(8):3073-6. doi: 10.1073/pnas.72.8.3073. PMID 810797
- [Background] Patrignani P, Filabozzi P, Patrono C. Selective cumulative inhibition of platelet thromboxane production by low-dose aspirin in healthy subjects. J Clin Invest. 1982 Jun;69(6):1366-72. doi: 10.1172/jci110576. PMID 7045161
- [Background] Reilly IA, FitzGerald GA. Inhibition of thromboxane formation in vivo and ex vivo: implications for therapy with platelet inhibitory drugs. Blood. 1987 Jan;69(1):180-6. PMID 3790723
- [Background] Mustard JF, Packham MA. The role of blood and platelets in atherosclerosis and the complications of atherosclerosis. Thromb Diath Haemorrh. 1975 Jun 30;33(3):444-56. PMID 1154306
- [Background] Mustard JF, Moore S, Packham MA, Kinlough-Rathbone RL. Platelets, thrombosis and atherosclerosis. Prog Biochem Pharmacol. 1977;13:312-25. PMID 928433
- [Background] Mustard JF, Packham MA, Kinlough-Rathbone RL. Platelets and thrombosis in the development of atherosclerosis and its complications. Adv Exp Med Biol. 1978;102:7-30. doi: 10.1007/978-1-4757-1217-9_2. No abstract available. PMID 356564
- [Background] Ikonomidis I, Andreotti F, Economou E, Stefanadis C, Toutouzas P, Nihoyannopoulos P. Increased proinflammatory cytokines in patients with chronic stable angina and their reduction by aspirin. Circulation. 1999 Aug 24;100(8):793-8. doi: 10.1161/01.cir.100.8.793. PMID 10458713
- [Background] Ridker PM, Cushman M, Stampfer MJ, Tracy RP, Hennekens CH. Inflammation, aspirin, and the risk of cardiovascular disease in apparently healthy men. N Engl J Med. 1997 Apr 3;336(14):973-9. doi: 10.1056/NEJM199704033361401. PMID 9077376
- [Background] Hennekens CH, Schror K, Weisman S, FitzGerald GA. Terms and conditions: semantic complexity and aspirin resistance. Circulation. 2004 Sep 21;110(12):1706-8. doi: 10.1161/01.CIR.0000142056.69970.DB. No abstract available. PMID 15381661
- [Background] Steer KA, Wallace TM, Bolton CH, Hartog M. Aspirin protects low density lipoprotein from oxidative modification. Heart. 1997 Apr;77(4):333-7. doi: 10.1136/hrt.77.4.333. PMID 9155612
- [Background] Wu R, Lamontagne D, de Champlain J. Antioxidative properties of acetylsalicylic Acid on vascular tissues from normotensive and spontaneously hypertensive rats. Circulation. 2002 Jan 22;105(3):387-92. doi: 10.1161/hc0302.102609. PMID 11804997
- [Background] Oberle S, Polte T, Abate A, Podhaisky HP, Schroder H. Aspirin increases ferritin synthesis in endothelial cells: a novel antioxidant pathway. Circ Res. 1998 May 18;82(9):1016-20. doi: 10.1161/01.res.82.9.1016. PMID 9598599
- [Background] Grosser N, Abate A, Oberle S, Vreman HJ, Dennery PA, Becker JC, Pohle T, Seidman DS, Schroder H. Heme oxygenase-1 induction may explain the antioxidant profile of aspirin. Biochem Biophys Res Commun. 2003 Sep 5;308(4):956-60. doi: 10.1016/s0006-291x(03)01504-3. PMID 12927812
- [Background] Hennekens CH, Dyken ML, Fuster V. Aspirin as a therapeutic agent in cardiovascular disease: a statement for healthcare professionals from the American Heart Association. Circulation. 1997 Oct 21;96(8):2751-3. doi: 10.1161/01.cir.96.8.2751. No abstract available. PMID 9355934
- [Background] U.S. Preventive Services Task Force. Aspirin for the primary prevention of cardiovascular events: recommendation and rationale. Ann Intern Med. 2002 Jan 15;136(2):157-60. doi: 10.7326/0003-4819-136-2-200201150-00015. PMID 11790071
- [Background] Hennekens CH, Hollar D, Baigent C. Sex-related differences in response to aspirin in cardiovascular disease: an untested hypothesis. Nat Clin Pract Cardiovasc Med. 2006 Jan;3(1):4-5. doi: 10.1038/ncpcardio0420. No abstract available. PMID 16391594
- [Background] Pearson TA, Blair SN, Daniels SR, Eckel RH, Fair JM, Fortmann SP, Franklin BA, Goldstein LB, Greenland P, Grundy SM, Hong Y, Miller NH, Lauer RM, Ockene IS, Sacco RL, Sallis JF Jr, Smith SC Jr, Stone NJ, Taubert KA. AHA Guidelines for Primary Prevention of Cardiovascular Disease and Stroke: 2002 Update: Consensus Panel Guide to Comprehensive Risk Reduction for Adult Patients Without Coronary or Other Atherosclerotic Vascular Diseases. American Heart Association Science Advisory and Coordinating Committee. Circulation. 2002 Jul 16;106(3):388-91. doi: 10.1161/01.cir.0000020190.45892.75. No abstract available. PMID 12119259

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From Dec 2006 through May 2007, 70 eligible subjects were randomized from a primary care clinical site under the direction of Alex Pokov, MD.
Pre-assignment Details: In this trial there was no wash-out or run-in period, as all eligible subjects were not taking aspirin.
Groups:
- Arm 1 of 5 Randomized Treatment Arms: 81 mg Aspirin
- Arm 2 of 5 Randomized Treatment Arms: 162 mg Aspirin
- Arm 3 of 5 Randomized Treatment Arms: 325 mg Aspirin
- Arm 4 of 5 Randomized Treatment Arms: 650 mg Aspirin
- Arm 5 of 5 Randomized Treatment Arms: 1300 mg Aspirin
Period: Overall Study
Arm/Group | Arm 1 of 5 Randomized Treatment Arms | Arm 2 of 5 Randomized Treatment Arms | Arm 3 of 5 Randomized Treatment Arms | Arm 4 of 5 Randomized Treatment Arms | Arm 5 of 5 Randomized Treatment Arms
Started | 14 | 14 | 14 | 14 | 14
Completed | 14 | 14 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 of 5 Randomized Treatment Arms | Arm 2 of 5 Randomized Treatment Arms | Arm 3 of 5 Randomized Treatment Arms | Arm 4 of 5 Randomized Treatment Arms | Arm 5 of 5 Randomized Treatment Arms | Total
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 11 | 11 | 8 | 51
  >=65 years | 3 | 4 | 3 | 3 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (10.3) | 57.0 (10.0) | 55.5 (9.2) | 58.0 (9.6) | 59.1 (11.4) | 57.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 5 | 5 | 9 | 33
  Male | 10 | 4 | 9 | 9 | 5 | 37
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 14 | 14 | 14 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Nitric Oxide Formation From Baseline to 3 Months
Description: Changes in Heme oxygenase (HO-1) a downstream target of nitric oxide (NO) formation.
Time Frame: Baseline to 3 Months (90-97 days)
Population: Complete baseline and follow-up data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1 of 5 Randomized Treatment Arms | Arm 2 of 5 Randomized Treatment Arms | Arm 3 of 5 Randomized Treatment Arms | Arm 4 of 5 Randomized Treatment Arms | Arm 5 of 5 Randomized Treatment Arms
Number analyzed (Participants) | 14 | 11 | 12 | 10 | 13
ng/mL | 27.6 (4.9) | 27.0 (4.4) | 31.4 (9.8) | 25.7 (3.4) | 28.3 (4.1)

2. Other Pre Specified Outcome: Change in Inflammatory Markers From Baseline to 3 Months.
Time Frame: Baseline to 3 Months (90-97 days)
Population: At the end of the study, due to lack of funds, analysis of this outcome was not conducted.
Arm/Group | Arm 1 of 5 Randomized Treatment Arms | Arm 2 of 5 Randomized Treatment Arms | Arm 3 of 5 Randomized Treatment Arms | Arm 4 of 5 Randomized Treatment Arms | Arm 5 of 5 Randomized Treatment Arms
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Other Pre Specified Outcome: Change in Platelet Biomarkers From Baseline to 3 Months.
Time Frame: Baseline to 3 Months (90-97 days)
Population: At the end of the study due to lack of funds analysis of this data was not conducted.
Arm/Group | Arm 1 of 5 Randomized Treatment Arms | Arm 2 of 5 Randomized Treatment Arms | Arm 3 of 5 Randomized Treatment Arms | Arm 4 of 5 Randomized Treatment Arms | Arm 5 of 5 Randomized Treatment Arms
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm 1 of 5 Randomized Treatment Arms | Arm 2 of 5 Randomized Treatment Arms | Arm 3 of 5 Randomized Treatment Arms | Arm 4 of 5 Randomized Treatment Arms | Arm 5 of 5 Randomized Treatment Arms
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No